CLINICAL TRIAL: NCT04997876
Title: Diagnostic Reliability of OCT Biomarkers for Idiopathic Epiretinal Membranes
Brief Title: Diagnostic Reliability of OCT Biomarkers for iERM
Status: Completed | Type: Observational
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Prof., MD, MBA, Vienna Institute for Research in Ocular Surgery
Other Study IDs: biomarkers
Record Dates: First submitted 2021-08-02; First posted 2021-08-10 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Idiopathic Epiretinal Membranes

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group: Biomarkers from presurgical OCTs are diagnosed
  Interventions: Other: Biomarker analysis

INTERVENTIONS:
Other: Biomarker analysis — Biomarkers from presurgical OCTs are assessed

SUMMARY:
Several optical coherence tomography (OCT) biomarkers with potential to influence postsurgical outcomes after vitrectomy with membrane peeling for idiopathic epiretinal membranes (iERM) have been described in single predictor analyses in the past. Aim of the study is to assess the reliability of diagnosis of OCT biomarkers and to calculate their impact on postsurgical visual acuity in a multiple regression analysis.

DETAILED DESCRIPTION:
Several optical coherence tomography (OCT) biomarkers with potential to influence postsurgical outcomes after vitrectomy with membrane peeling for idiopathic epiretinal membranes (iERM) have been described in single predictor analyses in the past. A recent multifactorial analysis outlined macular thickness and DRIL to be significant predictors for postsurgical visual acuity (Karasavviodou et al.). Nevertheless, reliability of diagnosing OCT biomarkes among patients with iERM was not yet assessed, to our knowledge. Aim of the study is to assess the reliability of diagnosis of OCT biomarkers and to calculate their impact on postsurgical visual acuity in a multiple regression analysis.

ELIGIBILITY:
Inclusion Criteria:

* a) presence of an iERM,
* b) indication for membrane peeling, defined as significant loss of visual acuity and/or metamorphopsia due to the ERM,
* c) pseudophakia at the final visit at 3 months after surgery, and
* d) written informed consent for study participation.

Exclusion Criteria:

* macular edema caused by conditions other than ERM were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with iERM sheduled for vitrectomy with membrane peeling.
Sampling Method: Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2021-08-05 (Actual); Study Completion 2021-08-21 (Actual)

PRIMARY OUTCOMES:
reliability of diagnosing OCT biomarkers | 1 week
  The presence (yes/no) of following OCT biomarkers are diagnosed from preoperative OCTs: EIFL, DRIL, intraretinal cystoid changes, alterations of the ellipsoid zone, cotton ball sign, HR-foci, EMM-rips, and retinal contraction. Intra- and interobserver reliability is assessed from 2 different readers, and reliability of OCT biomarkers will be calculated with the Kuder Richardson 20 test, due to the dichtomic nature of outcomes.

SECONDARY OUTCOMES:
postsurgical best corrected visual acuity | 3 months
  best corrected visual acuity 3 months after surgery is used for regression analysis
central macular thickness | 5 minutes
  presurgical central subfield thickness of the macula is assessed by the software of the OCT device. The subfield thickness with a diameter of 1mm will be selected.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Findl, Prof., Principal Investigator — head of department
Locations (1):
- VIROS at Hanusch-Hospital Vienna, Vienna, Austria

REFERENCES:
- [Background] Karasavvidou EM, Panos GD, Koronis S, Kozobolis VP, Tranos PG. Optical coherence tomography biomarkers for visual acuity in patients with idiopathic epiretinal membrane. Eur J Ophthalmol. 2021 Nov;31(6):3203-3213. doi: 10.1177/1120672120980951. Epub 2020 Dec 14. PMID 33307784